CLINICAL TRIAL: NCT04056481
Title: Expanded Access Protocol of Givosiran for Patients With Acute Hepatic Porphyria (AHP)
Brief Title: Expanded Access Protocol of Givosiran for Patients With Acute Hepatic Porphyria
Status: Approved for marketing | Type: Expanded Access
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-AS1-005
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Acute Hepatic Porphyria
Keywords: Acute Hepatic Porphyria (AHP); Acute Intermittent Porphyria (AIP); Porphyria; Acute Intermittent; Acute Porphyria; Hereditary Coproporphyria (HCP); Variegate Porphyria (VP); ALA Dehydratase Deficient Porphyria (ADP); Givosiran; Expanded Access; EAP
MeSH Terms: conditions — Coproporphyria, Hereditary; Porphyria, Acute Intermittent; Porphyrias; Porphyria, Variegate | interventions — givosiran

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Givosiran — givosiran (ALN-AS1) administered as a subcutaneous (SC) injection
  Other Names: ALN-AS1

SUMMARY:
The purpose of this study is to provide expanded access of givosiran to patients with Acute Hepatic Porphyria (AHP).

DETAILED DESCRIPTION:
Choosing to participate in an expanded access program is an important personal decision. Talk with your doctor and family members or friends about deciding to join a research study. To learn more about this study, please have your doctor contact the study research staff using the Contacts provided. For general information, see the link provided in More Information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Acute Hepatic Porphyria (Acute Intermittent Porphyria, Hereditary Coproporhyria, Variegate Porphyria, ALA dehydratase deficient porphyria)
* Have adequate venous access for program sample collections as judged by the Investigator for study sample collections

Exclusion Criteria:

* Previously or currently participating in a givosiran clinical trial
* Has any of the following laboratory parameter assessments at Screening:

  1. Alanine aminotransferase (ALT) >2×ULN
  2. Total bilirubin >1.5×ULN. Patients with elevated total bilirubin that is secondary to documented Gilbert's syndrome are eligible if the total bilirubin is <2×ULN
  3. Estimated Glomerular Filtration Rate (eGFR) <15 mL/min/1.73 m2
* On an active liver transplantation waiting list

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals